CLINICAL TRIAL: NCT02583477
Title: A Phase Ib and II Open-Label, Multi-Center Study of MEDI4736 Evaluated in Different Combinations in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Phase Ib/II Study of MEDI4736 Evaluated in Different Combinations in Metastatic Pancreatic Ductal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4198C00003
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma, PDAC, immunotherapy, PDL1, AZD5069, MEDI4736
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia | interventions — durvalumab; 130-nm albumin-bound paclitaxel; Gemcitabine; N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI4736 +nab-paclitaxel + gemcitabine (Experimental): MEDI4736 in combination with nab-paclitaxel + gemcitabine chemotherapy regimen via IV infusion
  Interventions: Drug: MEDI4736 in combination with nab-paclitaxel and gemcitabine
- MEDI4736+AZD5069 (Experimental): MEDI4736 via IV infusion and oral AZD5069
  Interventions: Drug: MEDI4736 in combination with AZD5069

INTERVENTIONS:
Drug: MEDI4736 in combination with nab-paclitaxel and gemcitabine — MEDI4736 in combination with nab-paclitaxel + gemcitabine chemotherapy regimen via IV infusion
  Arms: MEDI4736 +nab-paclitaxel + gemcitabine
Drug: MEDI4736 in combination with AZD5069 — MEDI4736 via IV infusion and oral AZD5069
  Arms: MEDI4736+AZD5069

SUMMARY:
A Phase Ib and II Open-Label, Multi-Center Study of MEDI4736 Evaluated in Different Combinations (with chemotherapy or AZD5069) in Patients with Metastatic Pancreatic Ductal Adenocarcinoma

DETAILED DESCRIPTION:
This is a Phase Ib and II open-label, multi-center study to evaluate the safety, tolerability, pharmacodynamics, and antitumor activity of MEDI4736 in combination with chemotherapy or AZD5069 in patients with pancreatic ductal adenocarcinoma (PDAC). This study will consist of 2 independent cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic PDAC, no more than 1 prior chemotherapy regimen or treatment-naïve patients
2. Eastern Cooperative Oncology Group 0 or 1
3. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) scan and that is suitable for accurate repeated measurements
4. MEDI4736 + nab-paclitaxel + gemcitabine chemotherapy cohort: treatment-naïve patients with metastatic PDAC who have received no previous systemic chemotherapy 5 MEDI4736 + Cohort: Patient should receive no more than 1 prior systemic chemotherapy regimen.

6. Life expectancy ≥ 12 weeks. 7. ECOG PS of 0 or 1 8. Adequate organ and bone marrow function 9. Ability to undergo during screening a tumor biopsy that is adequate for biomarker analysis.

Exclusion Criteria:

1. Any concurrent chemotherapy, investigational product , biologic, or hormonal therapy for cancer treatment.
2. Receipt of any investigational anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study treatment.
3. Major surgical procedure within 21 days prior to the first dose of IP.
4. Patients weighing less than 30 kg
5. History of leptomeningeal carcinomatosis
6. Ascites requiring intervention
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy
8. Current or prior use of immunosuppressive medication within 14 days of first dose
9. Brain metastases or spinal cord compression.
10. Medi4736+AZD5069 Cohort only: received any potent and moderate cytochrome CYP3A4 inhibitors, potent and moderate CYP3A4 inducers, P-gp substrates, BCRP substrates, sensitive CYP2B6 substrates, warfarin and coumarin derivatives, or herbal supplements within 14 days of the first dose of study treatment
11. Uncontrolled intercurrent illness
12. Other malignancy within 5 years except for noninvasive malignancies
13. Mean QT interval ≥470 ms
14. Active infection
15. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP
16. Female patients who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not employing an effective method of birth control
17. Prior exposure to immune-mediated therapy
18. Known allergy or hypersensitivity to IP formulations or to other human monoclonal antibodies

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Evans, M.D, Principal Investigator — Beatson Institute, University of Glasgow, Garscrube Estate, Switchback Rd. Glasgow, UK, G61 1BD
Locations (6):
- Research Site, Rochester, New York, United States
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral

REFERENCES:
- See also: CSP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3998&filename=d4198c00003-csp-v5-redact.pdf
- See also: SAP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3998&filename=d4198c00003-sap-ed-1-redact.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 independent cohorts, each of which ran at separate times between 25 March 2016 and 09 July 2018. In Cohort 1, participants were recruited from 1 center in the United States; in Cohort 2, participants were recruited from 6 centers in the United Kingdom.
Pre-assignment Details: Participants underwent screening evaluations to determine eligibility within 4 weeks (28 days) prior to first administration of the Investigational Product (IP). A total of 27 participants (3 in Cohort 1 and 24 in Cohort 2) were assigned to treatment and 23 were treated. Only treated participants are included in the participant flow.
Groups:
- Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine): Participants with metastatic pancreatic ductal adenocarcinoma (PDAC) who were treatment naive received MEDI4736 1.5 gram (g) intravenous (IV) infusion on Day 1 of each 28-day cycle (q4w). Participants also received nab-paclitaxel 125 milligram per meter square (mg/m^2) IV infusion followed by gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28-day cycle. Treatment continued until either confirmed progressive disease (PD) unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Cohort 2 (MEDI4736 + AZD5069): Participants with metastatic PDAC with progression on the indicated types of chemotherapy received MEDI4736 1.5 g IV infusion q4w. Participants also received AZD5069 orally twice daily (bid). The starting dose of 80 mg orally bid (with dose reductions to 40 mg or 20 mg for toxicity allowable). Treatment continued until either confirmed PD, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) | Cohort 2 (MEDI4736 + AZD5069)
Started | 3 | 20
Received Treatment | 3 | 20
Completed Treatment | 0 | 0
Completed (Completed study) | 0 | 0
Not Completed | 3 | 20
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 16
Not completed — Study terminated | 2 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of IP and for whom any post-dose data were available.
Groups:
- Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine): Participants with metastatic PDAC who were treatment naive received MEDI4736 1.5 g IV infusion q4w. Participants also received nab-paclitaxel 125 mg/m^2 IV infusion followed by gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28-day cycle. Treatment continued until either confirmed PD unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Cohort 2 (MEDI4736 + AZD5069): Participants with metastatic PDAC with progression on the indicated types of chemotherapy received MEDI4736 1.5 g IV infusion q4w. Participants also received AZD5069 orally bid. The starting dose of 80 mg orally bid (with dose reductions to 40 mg or 20 mg for toxicity allowable). Treatment continued until either confirmed PD, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) | Cohort 2 (MEDI4736 + AZD5069) | Total
Number analyzed (Participants) | 3 | 20 | 23
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 0 | 4 | 4
  >=50 - <65 years | 1 | 12 | 13
  >=65 - <75 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 1 | 11 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  White | 3 | 18 | 21
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT period was defined as first treatment cycle for Cohort 1, and first dose of AZD5069 and MEDI4736 to end of Cycle 1 or until a participant experienced a DLT, whichever occurs first for Cohort 2.
  A DLT was defined as any of below listed laboratory abnormalities or adverse events (AE) related to MEDI4736 collected during DLT period.
  * Liver transaminase elevation >= 5× but <= 8× upper limit of normal (ULN) that doesn't resolve to Grade 2 within 5 days
  * Transaminase elevation > 8× ULN or total bilirubin > 5× ULN
  * Any Grade 4 immune-related AE (irAE) not attributed to local tumor response, Grade >=3 colitis, Grade >=2 pneumonitis that doesn't resolve to <= Grade 1 within 7 days, Grade 3 irAE, that doesn't resolve to Grade <=1 or baseline status within 14 days
  * Any Grade >=3 non-irAE toxicity that doesn't resolve to Grade <=1 or baseline status within 14 days A DLT was defined as any Grade 3 or worse AE related to AZD5069 that occurs from first dose of AZD5069 up to end of DLT period.
Time Frame: Cohort 1: From time of first dose of MEDI4736 on Day 1 up to Day 28 of Cycle 1 and Cohort 2: From time of first dose of AZD5069 and MEDI4736 on Day 1 up to Day 28 of Cycle 1 or until a participant experiences a DLT, whichever occurs first.
Population: For Cohort 1: Participants who completed DLT evaluation period and/or discontinued study treatment early due to a DLT and who have not missed >=2 infusions of gemcitabine.
  For Cohort 2: Participants who received 50% of planned doses of AZD5069 during DLT period as well as MEDI4736 infusion and remained active on study at end of Day 28 of Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 3 | 12
Participants | 0 | 4

2. Primary Outcome: Number of Participants With AEs
Description: An AE is the development of an undesirable medical condition or deterioration of a pre-existing medical condition following or during exposure to study treatment, whether or not considered causally related to study treatment. An undesirable medical condition can be symptoms, signs or abnormal results of an investigation. A serious AE (SAE) is an AE that fulfills one or more following criteria: death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity or substantial disruption of ability to conduct normal life functions, congenital abnormality or birth defect, and an important medical event that may jeopardize participant or may require medical intervention to prevent one of outcomes listed above. AEs leading to discontinuation of study treatment were those with action taken was 'Drug Permanently Discontinued' for any study treatment. Only treatment emergent AEs were presented.
Time Frame: From first dose of study treatment administration (Day 1) until 90 days after the last dose of IP or initiation of the first subsequent anticancer therapy (whichever occurred first), approximately 30 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 3 | 20
Participants
  Any AE | 3 | 20
  Any AE causally related to treatment (CRT) | 3 | 14
  Any AE of CTCAE Grade 3 or higher | 3 | 18
  Any AE of CTCAE Grade 3 or higher CRT | 3 | 10
  Any AE leading discontinuation of study treatment | 2 | 3
  Any AE with outcome of death | 1 | 4
  Any AE with outcome of death CRT | 1 | 0
  Any SAE | 1 | 16
  Any SAE CRT | 1 | 8

3. Primary Outcome: Objective Response Rate (ORR) in Cohort 2
Description: ORR is defined as the percentage of participants with a confirmed overall response of complete response (CR) or partial response (PR). A confirmed response of CR/PR means that a response of CR/PR is recorded at 1 visit and confirmed by repeat imaging, preferably at the next regularly scheduled imaging visit and not less than 4 weeks after the visit when the response was first observed with no evidence of progression between the initial and CR/PR confirmation visit. CR is defined as disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters of TLs, taking as reference the baseline sum of diameters as long as criteria for PD were not met. ORR was determined using Investigator assessments according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1).
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study treatment), every 6 weeks +/-7 days for first 48 weeks, then every 12 weeks +/-7 days thereafter until confirmed objective disease progression. Up to approximately 30 months.
Population: The efficacy analysis set included all participants who received at least 1 dose of IP and with no important protocol deviation that could impact the efficacy evaluation.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
percentage of participants | 5.6 [0.58 to 19.95]

4. Secondary Outcome: Duration of Response (DoR) in Cohort 2
Description: DoR was defined as the time from the first documentation of CR/PR (which is subsequently confirmed) until the date of progression/death, or the last evaluable RECIST assessment for participants that did not progress or did progress after 2 missed visits of the last evaluable assessment (or first dose). PD was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. DoR was determined using Investigator assessments according to RECIST v1.1 and was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 3
Population: The efficacy analysis set included all participants who received at least 1 dose of IP and with no important protocol deviation that could impact the efficacy evaluation. Participants with confirmed response were evaluated, only one participant showed response.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 1
weeks | 18.29 [18.29 to 18.29]

5. Secondary Outcome: Disease Control Rate (DCR) in Cohort 2
Description: DCR at 6 months is defined as the percentage of participants who had a best objective response (BoR) of CR or PR in the first 6 months (i.e. 24+1=25 weeks to allow for a late assessment within the assessment window) or who had demonstrated stable disease (SD) for a minimum interval of 24 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e. 161 days) following the start of treatment. DCR at 12 months is defined as the percentage of participants who had a BoR of CR or PR in the first 12 months (i.e. 48+1=49 weeks to allow for a late assessment within the assessment window) or who had demonstrated SD for a minimum interval of 48 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e. 329 days) following the start of treatment. DCR was determined using Investigator assessments according to RECIST v1.1.
Time Frame: RECIST assessments were performed at baseline (within 28 days before start of study treatment) and every 6 weeks +/- 7 days for first 48 weeks up to 6 months and 12 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
percentage of participants
  At 6 months | 11.1
  At 12 months | 5.6

6. Secondary Outcome: Median Progression-Free Survival (PFS) in Cohort 2
Description: PFS is defined as the time from the date of first dose until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraws from allocated therapy or receives another anticancer therapy prior to progression. PFS was determined using Investigator assessments according to RECIST v1.1 and calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
months | 1.6 [1.29 to 1.68]

7. Secondary Outcome: Progression-Free Survival Rate at 3 Months (PFS3) in Cohort 2
Description: The PFS rate was defined as percentage of participants alive and progression-free after 3 months. The PFS3 was calculated using Kaplan-Meier estimates. Tumor progression was determined based on Investigator assessment and RECIST v1.1.
Time Frame: RECIST assessments were performed at baseline (within 28 days before start of study treatment) and every 6 weeks +/- 7 days up to 3 months
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
percentage of participants | 11.1 [3.91 to 22.55]

8. Secondary Outcome: Progression-Free Survival Rate at 6 Months (PFS6) in Cohort 2
Description: The PFS6 was defined as percentage of participants alive and progression-free after 6 months. The PFS6 was calculated using Kaplan-Meier estimates. Tumor progression was determined based on Investigator assessment and RECIST v1.1.
Time Frame: RECIST assessments were performed at baseline (within 28 days before start of study treatment) and every 6 weeks +/- 7 days up to 6 months
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
percentage of participants | 11.1 [3.91 to 22.55]

9. Secondary Outcome: Median Overall Survival (OS) in Cohort 2
Description: OS is defined as the time from the date of first dose until death due to any cause (i.e. date of death or censoring - date of first dose + 1). OS was calculated using the Kaplan-Meier technique. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive (censored at end of study).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
months | 2.8 [1.68 to 3.79]

10. Secondary Outcome: Overall Survival at 6 Months (OS6) in Cohort 2
Description: OS6 is defined as percentage of participants alive at 6 months from first dose of study treatment. OS6 was calculated using the Kaplan-Meier estimate of OS at 6 months.
Time Frame: From first dose of study treatment (Day 1) up to 6 months
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
percentage of participants | 22.2 [11.19 to 35.59]

11. Secondary Outcome: Overall Survival at 12 Months (OS12) in Cohort 2
Description: OS12 is defined as percentage of participants alive at 12 months from first dose of study treatment. OS12 was calculated using the Kaplan-Meier estimate of OS at 12 months.
Time Frame: From first dose of study treatment (Day 1) up to 12 months
Population: as for outcome 3
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 18
percentage of participants | 14.8 [5.74 to 27.92]

12. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADAs) for MEDI4736 in Cohort 2
Description: Samples were measured for the presence of ADAs and ADA-neutralizing antibodies for MEDI4736 using validated assays. Persistently positive is defined as positive at >=2 post-baseline assessments or positive at the last post-baseline assessment. Transiently positive is defined as having at least one post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive. NAB = neutralizing antibody.
Time Frame: On Day 1 of Cycles 1, 2, 3, 4, and 7; At months 3 and 6 after last dose
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 20
Participants
  Positive at any visit | 3
  Both baseline and post-baseline positive | 0
  Only post-baseline positive | 1
  Only baseline positive | 2
  ADA persistently positive | 0
  ADA transiently positive | 1
  ADA positive participants who are NAB positive | 0

13. Secondary Outcome: Mean Plasma Concentrations of MEDI4736 in Cohort 2
Description: Mean peak and trough plasma concentrations of MEDI4736 are presented.
Time Frame: Predose (within 60 minutes prior to treatment with any IP) on Day 1 of Cycles 1, 2, 3, 4, and 7; and post infusion (within 10 minutes after end of MEDI4736 infusion) on Day 1 of Cycles 1 and 7
Population: The Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of IP per protocol for whom any post-dose data were available and who did not violate or deviate from the protocol in ways that would significantly affect the PK analyses.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 20
nanograms per milliliter
  Cycle 1 Day 1: Predose: number analyzed (Participants) | 2
  Cycle 1 Day 1: Predose | 1444.730 (1010.7667)
  Cycle 1 Day 1: Post infusion | 339342.229 (95923.6405)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 11
  Cycle 2 Day 1: Predose | 56773.555 (17716.8788)
  Cycle 3 Day 1: Predose: number analyzed (Participants) | 6
  Cycle 3 Day 1: Predose | 63655.840 (26425.8402)
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 4
  Cycle 4 Day 1: Predose | 69325.233 (22750.3387)
  Cycle 7 Day 1: Predose: number analyzed (Participants) | 1
  Cycle 7 Day 1: Predose | 79687.820 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Cycle 7 Day 1: Post infusion: number analyzed (Participants) | 1
  Cycle 7 Day 1: Post infusion | 435297.610 (NA) — Standard deviation cannot be calculated when only one participant analyzed.

14. Secondary Outcome: Mean Plasma Concentrations of AZD5069 in Cohort 2
Description: Mean peak and trough plasma concentration of AZD5069 are presented. Concentration of AZD5069 was calculated by plasma concentration-time profile.
Time Frame: Predose (within 60 minutes prior to treatment with any IP) on Day 1 of Cycles 1, 2, 3, 4, and 7; and postdose (within 10 minutes after end of MEDI4736 infusion) on Day 1 of Cycles 1, 2, and 7
Population: The PK analysis set included all participants who received at least 1 dose of IP per protocol for whom any post-dose data were available and who did not violate or deviate from the protocol in ways that would significantly affect the PK analyses.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Cohort 2 (MEDI4736 + AZD5069)
Number analyzed (Participants) | 20
nanomoles per liter
  Cycle 1 Day 1: Predose | 10.60 (42.933)
  Cycle 1 Day 1: Postdose: number analyzed (Participants) | 19
  Cycle 1 Day 1: Postdose | 2236.29 (1678.496)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 11
  Cycle 2 Day 1: Predose | 1829.36 (1473.533)
  Cycle 2 Day 1: Postdose: number analyzed (Participants) | 1
  Cycle 2 Day 1: Postdose | 24.40 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Cycle 3 Day 1: Predose: number analyzed (Participants) | 5
  Cycle 3 Day 1: Predose | 502.48 (601.914)
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 4
  Cycle 4 Day 1: Predose | 1345.00 (1068.666)
  Cycle 7 Day 1: Predose: number analyzed (Participants) | 1
  Cycle 7 Day 1: Predose | 1200.00 (NA) — Standard deviation cannot be calculated when only one participant analyzed.
  Cycle 7 Day 1: Postdose: number analyzed (Participants) | 1
  Cycle 7 Day 1: Postdose | 7540.00 (NA) — Standard deviation cannot be calculated when only one participant analyzed.

ADVERSE EVENTS:
Time Frame: From initial IP administration (Day 1) until 90 days after the last dose of IP or initiation of the first subsequent anticancer therapy (whichever occurred first), approximately 30 months.
Description: The safety analysis set included all participants who received at least 1 dose of IP and for whom any post-dose data were available.
Arm/Group | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) | Cohort 2 (MEDI4736 + AZD5069)
All-Cause Mortality (participants affected / at risk) | 1/3 | 16/20
Serious Adverse Events (participants affected / at risk) | 1/3 | 16/20
Other Adverse Events (participants affected / at risk) | 3/3 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) (N=3) | Cohort 2 (MEDI4736 + AZD5069) (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (MEDI4736 + Nab-paclitaxel + Gemcitabine) (N=3) | Cohort 2 (MEDI4736 + AZD5069) (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Aptyalism (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (10)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 5 (5)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (10)
Administration site mass (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 10 (11)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 5 (5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (4)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (2)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Citrobacter test positive (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 7 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to a programmatic decision, enrollment of additional participants to cohort 1 was not pursued. The study was terminated by sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02583477/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT02583477/SAP_001.pdf